CLINICAL TRIAL: NCT01690091
Title: Cardioprotective and Metabolic Effects of Metformin in Patients With Heart Failure and Diabetes
Acronym: CARMET
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Terezie Pelikanova, Prof.MUDr.Terezie Pelikanova DrSc., Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NT13034
Record Dates: First submitted 2012-03-12; First posted 2012-09-21 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Insulin Resistance; Chronic Heart Failure
Keywords: chronic heart failure; type 2 diabetes; metformin; insulin resistance
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): 500 mg per day(1/2 tbl 1000 mg once a day - in the morning) after a week increase the dose to 1 tbl á 1000 mg after two weeks increase the dose to 2 x tbl 1000 mg (in the morning and in the evening), duration: 3 months
  Interventions: Drug: Metformini hydrochloridum (Siofor 1000 tbl, Berlin); Drug: placebo
- Placebo (Placebo Comparator): 500 mg per day(1/2 tbl 1000 mg once a day - in the morning) after a week increase the dose to 1 tbl á 1000 mg after two weeks increase the dose to 2 x tbl 1000 mg (in the morning and in the evening), duration:3 months
  Interventions: Drug: Metformini hydrochloridum (Siofor 1000 tbl, Berlin); Drug: placebo

INTERVENTIONS:
Drug: Metformini hydrochloridum (Siofor 1000 tbl, Berlin) — Patients will be randomized into 2 groups (A succession: MET-placebo, B succession: placebo-MET. After 3 months the treatment will be switched.
  Titration:
  500 mg per day(1/2 tbl 1000 mg once a day - in the morning) after a week increase the dose to 1 tbl á 1000 mg after two weeks increase the dose to 2 x tbl 1000 mg (in the morning and in the evening)
  Other Names: A10BA02 Metformin
Drug: placebo — Patients will be randomized into 2 groups (A succession: MET-placebo, B succession: placebo-MET. After 3 months the treatment will be switched.

SUMMARY:
The aim of the study is to evaluate the effect of metformin on myocardial function, insulin resistance and selected metabolic markers in patients with type 2 diabetes and heart failure (HF+DM+) in a cross-over, randomized, placebo controlled trial.

Hypothesis:

Metformin treatment in HF+DM+ group will lead to better myocardial function and load tolerance in comparison to placebo. The degree of improvement will be linked to selected metabolic parameters.

DETAILED DESCRIPTION:
40 patients with HF and DM without previous diabetes treatment will be randomized into 2 groups (A succession: MET-placebo, B succession: placebo-MET) - stratified randomization with following parameters weighted: HF etiology (ischemic /non-ischemic), diabetes duration, gender, BMI, age, NYHA, smoker/non-smoker). After 3 months the treatment will be switched. All participants will undergo standardized selection of metabolic and cardiovascular tests (hyperinsulinemic euglycemic clamp with indirect calorimetry, measurement of endothelial function, echocardiography, spiroergometry, proton/phosphor MR spectroscopy, adipose tissue biopsy, selected cytokines in plasma and adipose tissue at the beginning and the end of each intervention period (3 times in total).

ELIGIBILITY:
Inclusion Criteria:

1. chronic heart failure will be defined by the following criteria (all must be included):

   * diagnosis of HF known for at least 6 months
   * medical history of hospitalization for cardiac decompensation with need for parenteral therapy for congestion - X-ray findings or swelling of lower extremities
   * stable drug therapy at least 1 month
   * treatment with diuretics (thiazide or furosemide)
   * LVEF below 50%
2. the presence of diabetes will be defined by:

   * diagnosis and treatment of type 2 diabetes in the medical history
   * screening blood sample:

     * the value of HbA1c(according to IFCC)≥ 4.8% + fasting glucose ≥ 7.0 mmol / l in venous plasma or
     * the value of HbA1c ≥ 4.8%(according to IFCC) + random blood glucose ≥ 11.1 mmol/l in venous plasma
     * or OGTT - blood glucose level at 120 min ≥ 11.1 mmol/l OGTT is indicated just in case of positivity of one of the criteria (fasting glucose + HbA1c or HbA1c + random blood glucose)
   * treatment of diabetes - by diet only
   * women and men aged 40-70 years
   * body mass index (kg/m2) in the range of 20-35
   * the range of HbA1c between 4-6,5% IFCC
   * signed informed consent

Exclusion Criteria:

1. the planned cardiac intervention during the study that affect the function of the heart (revascularization including PCI, heart surgery, implantation of pacemaker, RF ablation; urgent candidate for OTS
2. metabolic disease, including: 1 type diabetes, decompensated thyreopathy (Note: patients with hypothyroidism and stable substitution (the last 3 months) of normal TSH levels may participate in the study
3. treatment with insulin or PAD one month before the recruitment(patients who were temporarily treated with insulin during hospitalization may participate in the study)
4. pregnancy (positive β-HCG test), breast feeding, trying to become pregnant
5. clinically significant anemia with hemoglobin below 100 g/l
6. renal insufficiency with eGF below 0.7 ml/s
7. atrial fibrillation - present during screening test
8. the presence of other medical condition, which occurs during physical examination, laboratory tests, ECG, including pulmonary, neurological or inflammatory disease, which would be considered by the examiner to distort the consistency of data

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | at baseline and after 3 months
  change of glucose disposal during clamp

SECONDARY OUTCOMES:
energy expenditure | at baseline and after 3 months
  change of energy expenditure measured by indirect calorimetry
endothelial function | at baseline and after 3 months
  change in digital pulse amplitude tonometry
heart function | at baseline and after 3 months
  change measured by echocardiography and spiroergometry

CONTACTS AND LOCATIONS:
Overall Officials: Terezie Pelikanova, Prof., MD, Principal Investigator — Diabetes Center, Institute of Clinical and Experimental Medicine
Locations (1):
- Diabetes Center, Institute of Clinical and Experimental Medicine, Prague, Czechia